CLINICAL TRIAL: NCT03801512
Title: Comparing the Efficacy of Transforaminal Epidural Injections, Acupuncture and Platelet Rich Plasma Injection in Patients with Sciatica Due to Intervertebral Disc Herniation, Spinal Stenosis and Spondylolisthesis
Brief Title: Comparing the Efficacy of Steroid, Acupuncture and Platelet Rich Plasma Injection in Patients with Sciatica
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Meng-Huang Wu, Attending physician, Department of Orthopedics, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201805024
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-04

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Steroids; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Steroid Injections (Experimental): Inject steroid at neuritis nerve root.
  Interventions: Other: Steroid
- Acupuncture (Experimental): Acupuncture at acupoints BL23 to BL26.
  Interventions: Other: Acupuncture
- Platelet Rich Plasma Injection (Experimental): Inject Platelet Rich Plasma at neuritis nerve root.
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Other: Steroid — Triamcinolone 1pc + lidocaine 1% 1cc inject at neuritis nerve roots
  Arms: Steroid Injections
Other: Acupuncture — 1.5 inch acupuncture needles insert at acupoints BL23, BL24, BL25 and BL26
  Arms: Acupuncture
Other: Platelet Rich Plasma — Inject investigators Platelet Rich Plasma at neuritis nerve roots
  Arms: Platelet Rich Plasma Injection

SUMMARY:
Disc herniation, stenosis of the spine and spondylolisthesis are the common causes of radiculitis in medical practice today, and can cause symptoms of sciatica. Steroid injection, acupuncture and platelet-rich plasma injection are often used interventions for the treatments of sciatica. The investigators will investigate the efficacy and safety of steroid injection, acupuncture and platelet-rich plasma injection for sciatica in this single center, parallel, randomized-controlled clinical trial.

DETAILED DESCRIPTION:
Steroid injection, acupuncture and platelet-rich plasma injection are often used interventions for the treatments of sciatica. The investigators will investigate the efficacy and safety of steroid injection, acupuncture and platelet-rich plasma injection for sciatica in this single center, parallel, randomized-controlled clinical trial.

Participants will be randomized into 3 groups (steroid injection, acupuncture and platelet-rich plasma injection) by central allocation. Randomized participants will complete a questionnaire that solicited information regarding age, sex, marital status, occupation, education, and medical history. The blinding credibility of the treatments will be evaluated at the end of the treatment.

Participants in steroid injection group will receive Triamcinolone 1pc plus lidocaine 1% 1cc injection at neuritis nerve roots. Participants in platelet-rich plasma injection group will receive 15cc blood draw first to concentrate into platelet-rich plasma and then inject at neuritis nerve roots. Participants in acupuncture group received standardized acupuncture treatment. hat treatment was accomplished by selecting a group of acupuncture points that predefined. Acupuncture points will be bladder meridian pattern acupuncture points including Shenshu (BL23), Qihaishu (BL24), Dachangshu (BL25), and Guanyuanshu(BL26). The needles will be inserted perpendicular to a depth of 5 to 35 mm depending on the acupuncture point, which was followed by manual stimulation by bidirectional rotation to induce Deqi sensation. Deqi was defined as a dull, localized, and aching sensation, which signaled the attainment of qi.

Outcome Measures Primary Outcome Measure The primary outcome measure is visual analogue scale for sciatica. To understand the impact of sciatica on the participants' life, visual analogue scale for bothersomeness is chosen instead of pain intensity. The participants will be asked to mark, on a 10 cm visual analogue scale (0, absence of bothersomeness; 10, the worst bothersomeness imaginable), the average degree of bothersomeness due to sciatica experienced within the most recent 1 week from the day of the assessment. This measurement has substantial validity. Bothersomeness of sciatica will be measured at baseline, 1-, 2-, 4-, 8-, 12-, 16-, and 24-week.

Secondary Outcome Measures Numeric Rating Scale for pain intensity is a simple method evaluating the subjective intensity of pain. Pain intensity will be measured in the same way as visual analogue scale for bothersomeness. Validity of its reliability has been demonstrated. The Chinese version Oswestry Disability Index is used to measure back pain-related dysfunction. Health-related quality of life will be measured using the well-validated EuroQol 5 dimensions (EQ-5D). A higher score is indicative of a better general health status. Participants satisfaction will be evaluated with 5 point scale (1 is worst, and 5 is best)

We will perform the Shapiro-Wilk normality test to determine whether or not the sample values followed a normal distribution and finally assumed normality according to the test result. For the description of baseline characteristics, mean with standard deviation (SD) for continuous data and frequency with percentage for dichotomous data will be described. Also, for the homogeneity test of baseline characteristics between 3 groups, 2-sample t tests for continuous data and chi-square test for dichotomous data will be performed. A mixed-model approach of repeated-measures 2-factor analysis will be used to analyze the difference and mean change in baseline, 1-, 2-, 4-, 8-, 12-, 16-, and 24-week visual analogue scale score, Oswestry Disability Index, EQ-5D, patient satisfaction difference and mean change between groups, interaction between groups, and periods.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, 20 to 80 years of age.
2. Participants who had dermatome between L3 to S1, or participants whose straight leg raising test was positive, or participants had Meyerding Grade I to II spondylolisthesis or herniated intervertebral disc or spinal stenosis diagnosed by X-rays, Magnetic resonance imaging or computed tomography.
3. Participants whose sciatica symptom doesn't have occur time limit.
4. Participants who agreed to follow the trial protocol.
5. Participants who could complete the study treatment and assessments.
6. Participants who had steroid or pain control injection can participate the study after receiving injection more than 3 days.

Exclusion Criteria:

1. Participants with severe progressive neurological symptoms (e.g. cauda equina compression).
2. Participants who had undergone surgery for lumbar disc herniation within 6 months.
3. Participants whose sciatica symptom wasn't caused by lumbar radiculopathy.
4. Participants with cardiovascular, liver, kidney, or hematopoietic system diseases, severe psychiatric or psychological disorder, or cancer.
5. Women who were pregnant.
6. Participants with a pacemaker, metal allergy, or severe fear of needles.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale score | 2 weeks
  Self reported pain intensity: 1. scales with a middle point, graduations or numbers; 2. meter-shaped scales; 3. "box-scales" consisting of circles equidistant from each other; 4. scales with descriptive terms at intervals along a line

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | 2 weeks
  An 11-point scale for patient self-reporting of pain scored 0-10 ( 0=no pain, 10= pain as bad as can be)
EQ-5D | 2 weeks
  The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are.
Oswestry Disability Index (ODQ) | 2 weeks
  The Oswestry Disability Index (ODQ) has ten sections: pain, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and travelling. Respondents choose one of six statements that most applies to them in each section. The first statement is scored 0, the second is scored 1, and so on to 5 for the sixth statement. The sum of the section scores is transformed to a percentage score, adjusted for missed sections. The total possible score ranges 0-100 and a higher score indicates worse function. Scores from 0-20% are claimed to indicate 'minimal disability', 20-40% 'moderate disability', 40-60% 'severe disability', 60-80% 'crippled', and 80-100% 'bedbound or exaggerating'

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Jade Chen, PhD, Study Chair — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Inoue M, Hojo T, Yano T, Katsumi Y. Electroacupuncture direct to spinal nerves as an alternative to selective spinal nerve block in patients with radicular sciatica--a cohort study. Acupunct Med. 2005 Mar;23(1):27-30. doi: 10.1136/aim.23.1.27. PMID 15844437
- [Background] Abbasipour-Dalivand S, Mohammadi R, Mohammadi V. Effects of Local Administration of Platelet Rich Plasma on Functional Recovery after Bridging Sciatic Nerve Defect Using Silicone Rubber Chamber; An Experimental Study. Bull Emerg Trauma. 2015 Jan;3(1):1-7. PMID 27162893
- [Background] Kucuk L, Gunay H, Erbas O, Kucuk U, Atamaz F, Coskunol E. Effects of platelet-rich plasma on nerve regeneration in a rat model. Acta Orthop Traumatol Turc. 2014;48(4):449-54. doi: 10.3944/AOTT.2014.13.0029. PMID 25230270
- [Background] Centeno C, Markle J, Dodson E, Stemper I, Hyzy M, Williams C, Freeman M. The use of lumbar epidural injection of platelet lysate for treatment of radicular pain. J Exp Orthop. 2017 Nov 25;4(1):38. doi: 10.1186/s40634-017-0113-5. PMID 29177632